CLINICAL TRIAL: NCT03818659
Title: Improving Blood Pressure Control in Diverse Populations by Measuring Accurately, Acting Rapidly, and Partnering With Patients
Brief Title: Improving BP Control in Diverse Populations Using BP MAP
Acronym: BP MAP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: OCHIN, Inc. (Other); Louisiana Public Health Institute (Other); American Medical Association (Other); American Heart Association (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 18-25890
Record Dates: First submitted 2019-01-22; First posted 2019-01-28 (Actual); Results first posted 2025-03-03 (Actual); Last update posted 2025-03-03 (Actual); Status verified 2025-02

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Self-Guided (Active Comparator): Active Clinics randomized to the Self-Guided Arm will receive access to an AHA/AMA web platform that includes the posted M.A.P. materials and limited access to AMA Staff who are available to answer questions. The study team will facilitate access to staff by hosting a kick-off webinar for program participants that will include an orientation to the materials on the website, general advice and practical tips about what works for implementation, and time for answering questions and discussion with the group.
  Interventions: Other: Self-Guided M.A.P. BP Improvement Program
- Full Support (Experimental): Active Clinics randomized to the Full Support Arm will receive online access to M.A.P. materials and orientation webinar and also a Practice Change Facilitator who will lead the health center clinical staff, site champions and physician leads at each clinic over the course of 6 months to support the implementation of the MAP Program. With support from an AMA "Improvement Advisor", the Practice Change Facilitators will perform a baseline assessment of current workflows and assess each domain of M.A.P. The goal of the Full Support program is to help care teams develop skills and sustainable workflows that are effective at attaining and maintaining high levels of BP control.
  Interventions: Other: Full Support M.A.P. BP Improvement Program
- Usual Care (No Intervention): The investigators will also conduct non-randomized comparisons of BP control in the Full Support and Self-Guided intervention arms to BP control in non-participating "Usual Care" institutions in PCORnet.

INTERVENTIONS:
Other: Self-Guided M.A.P. BP Improvement Program — Active Clinics randomized to the Self-Guided Arm will receive access to an AHA/AMA web platform that includes the posted M.A.P. materials and limited access to AMA Staff who are available to answer questions. The study team will facilitate access to staff by hosting a kick-off webinar for program participants that will include an orientation to the materials on the website, general advice and practical tips about what works for implementation, and time for answering questions and discussion with the group.
  Arms: Self-Guided
Other: Full Support M.A.P. BP Improvement Program — Active Clinics randomized to the Full Support Arm will receive online access to M.A.P. materials and orientation webinar and also a Practice Change Facilitator who will lead the health center clinical staff, site champions and physician leads at each clinic over the course of 6 months to support the implementation of the MAP Program. With support from an AMA "Improvement Advisor", the Practice Change Facilitators will perform a baseline assessment of current workflows and assess each domain of M.A.P. The goal of the Full Support program is to help care teams develop skills and sustainable workflows that are effective at attaining and maintaining high levels of BP control.
  Arms: Full Support

SUMMARY:
BP-MAP is a cluster randomized controlled trial (RCT) designed to compare the effectiveness of BP lowering from a clinic-based quality improvement program with Full Support (dedicated practice facilitation) vs. a Self-Guided version of the program. The American Medical Association (AMA) developed the framework for the interventions.

DETAILED DESCRIPTION:
BP-MAP is a cluster randomized controlled trial (RCT) designed to compare the effectiveness of BP lowering from a clinic-based quality improvement program with Full Support (dedicated practice facilitation) vs. a Self-Guided version of the program. The American Medical Association (AMA) developed the framework for the interventions. The trial will be conducted within the National Patient-Centered Clinical Research Network (PCORnet) that enables distributed querying of electronic health record data in a common data model. The primary outcome will be change in clinic-level blood pressure (BP) control at 6 months. Secondary outcomes will include other blood pressure (BP) control metrics, other time points (12 and 18 months), and process measures such as BP measurement accuracy, medication intensification, and average systolic blood pressure (SBP) reduction after a medication intensification, and repeat visit within 4 weeks after a visit with elevated BP. The investigators hypothesize clinics randomized to the Full Support version will achieve a larger increase from baseline in the proportion of their hypertensive patients with controlled BP at 6 months as compared to clinics randomized to the Self-Guided version, and also as compared with usual care. The investigators will also conduct non-randomized comparisons of BP control in the Full Support and Self-Guided intervention arms to BP control in non-participating "Usual Care" institutions in PCORnet. This study was submitted to the IRB at UCSF, determined to be quality improvement and exempt from further review.

ELIGIBILITY:
ACTIVE CLINICS

For inclusion as an Active Clinic in this study, clinics may participate must be able to identify:

* A Site Champion who works at the clinic and who is willing to take primary responsibility for implementing the M.A.P. intervention
* A Physician Champion who works at the clinic and who is willing to advocate actively for the M.A.P. intervention
* A Practice Change Facilitator willing to attend a 1-day training and help guide implementation of the M.A.P intervention for Full Support sites, with the support of AMA staff (may be the Site Champion or Physician Champion, or a person with regional responsibilities who can support multiple sites)

Sites will be excluded if they:

* Have implemented any high blood pressure quality improvement component from the M.A.P. BP improvement program as part of Target: BP or from the AMA or Target: BP websites
* Are currently involved in an ongoing clinical trial or grant funded project related to high blood pressure or hypertension

USUAL CARE CLINICS:

Usual Care Clinics will include PCORnet Datamarts participating in BP TRACK, a concurrently-running BP Control Registry within PCORnet that will provide quarterly datamart-level estimates of BP control and other aggregate metrics relevant to BP control. All participating datamarts will be included, with the following exceptions:

* Datamarts with any Active Clinics participating in BP MAP will be excluded
* Datamarts that obscure dates via date-shifting will be excluded, as this will not allow for control of concurrent secular trends

PATIENTS

Within clinics (Active or Usual Care), patients will be eligible (and identified from the electronic health record) if they meet National Quality Forum BP Control Metric (NQF 0018) criteria:

* Age 18-85 on the date of analysis
* At least one outpatient encounter with a diagnosis of hypertension during the first six months of the measurement year (ending on the date of analysis)
* No diagnosis or evidence of end-stage renal disease on or prior to the end of the measurement year
* No pregnancy during the measurement year
* No admission to an inpatient setting during the measurement year

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1238835 (Actual)
Dates: Start 2019-07-01 (Actual); Primary Completion 2021-02-28 (Actual); Study Completion 2021-06-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mark Pletcher, MD, MPH, Principal Investigator — University of California, San Francisco
Locations (24):
- United States (24):
  - Open Door Del Norte CHC, Crescent City, California
  - Open Door Eureka Community Health & Wellness Center, Eureka, California
  - QueensCare Echo Park Clinic, Los Angeles, California
  - Monterey County Health Department Laurel Family Practice, Salinas, California
  - Belle Chasse Community Health Center, Belle Chasse, Louisiana
  - Daughters of Charity Carrollton, Carrollton, Louisiana
  - St. Bernard Community Health Center, Chalmette, Louisiana
  - Daughters of Charity Gretna, Gretna, Louisiana
  - Daughters of Charity Kenner, Kenner, Louisiana
  - Kenner Community Health Center, Kenner, Louisiana
  - St Charles Community Health Center- Paul Maillard, Luling, Louisiana
  - St. Charles Community Health Center, Luling, Louisiana
  - Daughters of Charity Metairie, Metairie, Louisiana
  - Daughters of Charity St. Cecilia, New Orleans, Louisiana
  - Daughters of Charity Higgins, New Orleans, Louisiana
  - Daughters of Charity New Orleans East, New Orleans, Louisiana
  - Access Health Louisiana Primary Care at the Pythian, New Orleans, Louisiana
  - Daughters of Charity Gentilly, New Orleans, Louisiana
  - Waterfall CHC, North Bend, Oregon
  - Tillamook CHC, Tillamook, Oregon
  - Public Health: Seattle & King County Eastgate Public Health Center, Bellevue, Washington
  - Public Health: Seattle & King County Primary Care at Navos, Burien, Washington
  - Cowlitz County Health Department Cowlitz County: North Beach Clinic, Longview, Washington
  - Public Health: Seattle & King County Downtown Public Health Center, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Fontil V, Modrow MF, Cooper-DeHoff RM, Wozniak G, Rakotz M, Todd J, Azar K, Murakami L, Sanders M, Chamberlain AM, O'Brien E, Lee A, Carton T, Pletcher MJ. Improvement in Blood Pressure Control in Safety Net Clinics Receiving 2 Versions of a Scalable Quality Improvement Intervention: BP MAP A Pragmatic Cluster Randomized Trial. J Am Heart Assoc. 2023 Feb 7;12(3):e024975. doi: 10.1161/JAHA.121.024975. Epub 2023 Jan 25. PMID 36695297

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The unit of randomization was the participating clinical unit.
Pre-assignment Details: 24 clinic leaders agreed to participate in a BP control quality improvement program and 24 clinics were randomized and assigned to one of the intervention arms. We included 18 PCORnet clinics in our Blood Pressure Control Laboratory Surveillance Program (BP Track) for our control arms.
  No individuals were consented. This study was exempt from IRB review as a quality improvement program not human subjects research.
Units Other Than Participants: Number of clinic
Period: Overall Study
Arm/Group | Full Support | Self-Guided | Usual Care
Started | 11821; 12 Number of clinic (We had 10445 participants at baseline. Since we cannot report a greater number of participants that Completed the Period than the number of participants that Started the Period, we are reporting the Completed number.) | 14454; 12 Number of clinic (We had 13163 participants at baseline. Since we cannot report a greater number of participants that Completed the Period than the number of participants that Started the Period, we are reporting the Completed number.) | 1212560; 18 Number of clinic (We had 1177804 participants at baseline. Since we cannot report a greater number of participants that Completed the Period than the number of participants that Started the Period, we are reporting the Completed number.)
Completed | 11821; 12 Number of clinic | 14454; 12 Number of clinic | 1212560; 18 Number of clinic
Not Completed | 0; 0 Number of clinic | 0; 0 Number of clinic | 0; 0 Number of clinic

BASELINE CHARACTERISTICS:
Population: The unit of measure in this study is a clinic.
Units Other Than Participants: Number of Clinics
Groups:
- Total: Total of all reporting groups
Arm/Group | Full Support | Self-Guided | Usual Care | Total
Number analyzed (Participants) | 11821 | 14454 | 1212560 | 1238835
Number analyzed (Number of Clinics) | 12 | 12 | 18 | 42
Age, Continuous [Mean (Standard Deviation); unit: Age in years] | 57.1 (2.49) | 57.1 (2.61) | 63.47 (1.76) | 63.46 (1.78)
Age, Customized [Mean (Standard Deviation); unit: percentage of participants]
  18-44 years | 16.0 (4.91) | 16.1 (5.33) | 9.3 (2.21) | 13.8 (5.42)
  45-64 years | 56.5 (4.50) | 56.5 (6.07) | 38.1 (4.58) | 50.4 (10.06)
  65+ years | 27.5 (8.03) | 27.4 (8.38) | 52.6 (6.14) | 35.8 (14.09)
Sex/Gender, Customized [Mean (Standard Deviation); unit: percentage of participants]
  Female, % | 57.2 (5.80) | 60.7 (5.75) | 51.4 (3.08) | 56.4 (6.35)
  Male, % | 42.8 (5.80) | 39.3 (5.75) | 48.6 (3.08) | 43.6 (6.35)
Race/Ethnicity, Customized [Mean (Standard Deviation); unit: percentage of participants]
  White, % | 50.3 (33.8) | 29.8 (27.01) | 79.2 (15.56) | 53.1 (33.40)
  LatinX, % | 10.3 (5.9) | 26.3 (28.3) | 3.1 (2.01) | 13.2 (19.36)
  Black, % | 34.9 (33.8) | 36.8 (34.6) | 13.4 (15.3) | 28.4 (31.12)
  Asian, % | 1.6 (2.34) | 3.8 (5.69) | 1.7 (0.67) | 2.3 (3.72)
  Other, % | 3.0 (2.29) | 3.2 (2.69) | 2.5 (0.95) | 2.9 (2.14)
Median total number of patients with hypertension [Median (Inter-Quartile Range); unit: number of participants] | 517 [299 to 1049] | 1040 [630 to 1623] | 53266 [26200 to 74379] | 2003 [596 to 46407]
Diabetes, % [Mean (Standard Deviation); unit: percentage of participants] | 29.9 (3.43) | 33.8 (9.89) | 26.7 (2.74) | 26.7 (2.78)
Heart Failure, % [Mean (Standard Deviation); unit: percentage of participants] | 2.9 (1.51) | 2.6 (1.36) | 6.8 (1.30) | 6.8 (1.31)
Depression, % [Mean (Standard Deviation); unit: percentage of participants] | 17.0 (9.47) | 18.2 (16.4) | 14.5 (5.80) | 14.5 (5.83)
COPD (%) [Mean (Standard Deviation); unit: percentage of participants] | 6.6 (4.18) | 4.4 (2.43) | 5.7 (1.51) | 5.7 (1.51)

OUTCOME MEASURES:

1. Primary Outcome: Change in Blood Pressure Control, % of Patients
Description: The primary outcome will be clinic-level change in the proportion of patients with controlled BP from baseline to 6 months after the start of the intervention. BP control will be defined according to NQF 0018 as the percent of eligible patients (defined below) with SBP <140 mmHg and DBP < 90 mmHg, based on measurements obtained at the most recent ambulatory clinical encounter at baseline (using the lowest measures of SBP and DBP at that encounter) and similarly at the 6-month time point after initiation of the intervention.
Time Frame: baseline and 6 months
Population: The unit of measure in this study is a clinic. All patients with hypertension at each of the included clinics were analyzed and used to evaluate the numerator and denominator for each metric.
Measure: Mean (95% Confidence Interval); unit: percentage of patients
Units Other Than Participants: Number of Clinics
Arm/Group | Full Support | Self-Guided | Usual Care
Number analyzed (Participants) | 11821 | 14454 | 1212560
Number analyzed (Number of Clinics) | 12 | 12 | 18
percentage of patients | 2.8 [-0.9 to 6.5] | 1.6 [-0.8 to 4.0] | -0.4 [-1.0 to 0.2]

2. Secondary Outcome: Change in Improvement in Blood Pressure, % of Patients
Description: This overall measure of BP improvement implements CMS065v4[ref], which defines BP improvement as either a reduction of 10 mmHg in SBP or achievement of SBP that is "adequately controlled" (SBP < 140 mmHg) in months 12 of the measurement period, among hypertensive patients not previously controlled.
Time Frame: baseline and 12 months
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: percentage of patients
Units Other Than Participants: Number of Clinics
Arm/Group | Full Support | Self-Guided | Usual Care
Number analyzed (Participants) | 11821 | 14454 | 1212560
Number analyzed (Number of Clinics) | 12 | 12 | 18
percentage of patients | -3.4 [-10.3 to 3.5] | -5.4 [-8.2 to -2.5] | -3.1 [-4.1 to -2.1]

3. Secondary Outcome: Change in Confirmatory Repeated Blood Pressure Measurement, % of Visits
Description: This process measure is designed to capture the practice of repeating a blood pressure measurement in the same visit when the first measurement done in clinic is high (SBP≥140 mmHg or DBP≥90 mmHg).
Time Frame: baseline and 6 months
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: percentage of visits
Units Other Than Participants: Number of Clinics
Arm/Group | Full Support | Self-Guided | Usual Care
Number analyzed (Participants) | 11821 | 14454 | 1212560
Number analyzed (Number of Clinics) | 12 | 12 | 18
percentage of visits | 19.8 [6.9 to 32.7] | 11.6 [2.1 to 21.1] | 0.1 [-0.0 to 0.2]

4. Secondary Outcome: Change in Medication Intensification, % of Visits
Description: This process measure captures the proportion of visits where BP is uncontrolled where a medication is ordered that is of a different class of medication than had previously been used. Note that this explicitly does not give credit for ordering a simple refill or medication dose increase, or use of a different medication in the same class.
Time Frame: baseline and 6 months
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: percentage of visits
Units Other Than Participants: Number of Clinics
Arm/Group | Full Support | Self-Guided | Usual Care
Number analyzed (Participants) | 11821 | 14454 | 1212560
Number analyzed (Number of Clinics) | 12 | 12 | 18
percentage of visits | -1.6 [-6.1 to 3.0] | -3.4 [-8.2 to 1.2] | -0.1 [-0.3 to 0.1]

5. Secondary Outcome: Change in Average Systolic Blood Pressure (SBP) Reduction After a Medication Intensification Visit, mmHg
Description: This continuous metric describes the change in SBP (+/- standard deviation) observed between a visit with a medication intensification to the subsequent visit occurring at least 10 days later.
Time Frame: baseline and 6 months
Population: The unit of measure in this study is a clinic. All patients with hypertension at each of the included clinics were analyzed and used to evaluate the average reduction in patients with a recent medication intensification.
Measure: Mean (95% Confidence Interval); unit: mmHg
Units Other Than Participants: Number of Clinics
Arm/Group | Full Support | Self-Guided | Usual Care
Number analyzed (Participants) | 11821 | 14454 | 1212560
Number analyzed (Number of Clinics) | 12 | 12 | 18
mmHg | 2.3 [0.9 to 3.7] | -1.6 [-5.6 to 2.4] | -1.1 [-1.5 to -0.8]

6. Secondary Outcome: Change in Repeat Visit in 4 Weeks After a Visit With Elevated BP, % of Visits
Description: This process measure captures the proportion of persons who had uncontrolled HTN who made a subsequent visit within the following 4 weeks.
Time Frame: baseline and 6 months
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: percentage of visits
Units Other Than Participants: Number of Clinics
Arm/Group | Full Support | Self-Guided | Usual Care
Number analyzed (Participants) | 11821 | 14454 | 1212560
Number analyzed (Number of Clinics) | 12 | 12 | 18
percentage of visits | -0.8 [-3.2 to 1.7] | -2.0 [-4.3 to 0.2] | -0.6 [-1.0 to -0.2]

7. Secondary Outcome: Change in Use of Fixed Dose Combination Product Among Patients Taking 2 or More Classes of Medications, % of Patients
Description: Use of fixed dose combination medications helps with adherence, promotes rational combinations of medications, and increases likelihood of achieving BP control. This metric, which is limited to patients taking more than one medication class, describes the prevalence of fixed dose combination pill use.
Time Frame: baseline and 6 months
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: percentage of patients
Units Other Than Participants: Number of Clinics
Arm/Group | Full Support | Self-Guided | Usual Care
Number analyzed (Participants) | 11821 | 14454 | 1212560
Number analyzed (Number of Clinics) | 12 | 12 | 18
percentage of patients | 1.6 [-1.4 to 4.7] | -0.1 [-1.8 to 1.7] | -0.7 [-0.8 to -0.6]

8. Secondary Outcome: Change in Use of a CCB or Thiazide or Thiazide-like Diuretic Among African-American Patients on at Least One Medication, % of Patients
Description: Use of calcium channel blockers (CCB) OR a thiazide or thiazide-like diuretic medication classes is recommended to treat black or African American patients as first line monotherapy due to increased efficacy. This metric, which is limited to African-American patients with a diagnosis of hypertension taking at least one medication class, describes the prevalence of those receiving the recommended drug class.
Time Frame: baseline and 6 months
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: percentage of patients
Units Other Than Participants: Number of Clinics
Arm/Group | Full Support | Self-Guided | Usual Care
Number analyzed (Participants) | 11821 | 14454 | 1212560
Number analyzed (Number of Clinics) | 12 | 12 | 18
percentage of patients | -0.9 [-1.8 to 0.1] | -0.1 [-1.5 to 1.2] | 0.0 [-0.3 to 0.3]

9. Secondary Outcome: Change in Terminal Digit = Zero, % of Measurements
Description: Inappropriate rounding of blood pressure measurements (usually to zero) leads to measurement error and worse treatment decisions. This continuous metric is calculated for a clinic as the percent of measurements at that clinic (for hypertensive patients) where the terminal digit of the measurement is zero. A percent greater than 10% (if an automated BP monitor is used) or greater than 20% (if a manual BP monitor is used with recommended rounding to even digits) indicates evidence of inappropriate rounding. Unlike most of our metrics, lower is better, down to an ideal value of 10-20%, which would be expected if no rounding were occurring.
  For this study we calculated the change in this continuous metric for each clinic from baseline to 6 months, and then described the mean change across clinics by group. As with our other outcomes, the unit of analysis in the study is a clinic.
Time Frame: baseline and 6 months
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: percentage of measurements
Units Other Than Participants: Number of Clinics
Arm/Group | Full Support | Self-Guided | Usual Care
Number analyzed (Participants) | 11821 | 14454 | 1212560
Number analyzed (Number of Clinics) | 12 | 12 | 18
percentage of measurements | 0.8 [-1.5 to 3.1] | 0.9 [-1.1 to 2.8] | -0.6 [-1.0 to -0.3]

10. Secondary Outcome: Change in Blood Pressure Controlled to 2017 Guideline Goal, % of Patients
Description: This alternative overall measure of BP control is identical to Metric 1, except that attainment of BP Control is defined by SBP < 130 mmHg and DBP < 80 mmHg, as per the goal stated in the 2017 ACC/AHA Hypertension Guideline[ref]. Note that while the treatment threshold varies in the Guideline, depending on cardiovascular risk, the goal applies to all patients.
Time Frame: baseline and 6 months
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: percentage of patients
Units Other Than Participants: Number of clinic
Arm/Group | Full Support | Self-Guided | Usual Care
Number analyzed (Participants) | 11821 | 14454 | 1212560
Number analyzed (Number of clinic) | 12 | 12 | 18
percentage of patients | -1.5 [-2.6 to -0.3] | -1.1 [-2.2 to 0.1] | -0.5 [-0.7 to -0.2]

ADVERSE EVENTS:
Time Frame: Not applicable: adverse events were not collected.
Description: Adverse events were not collected.
Arm/Group | Full Support | Self-Guided | Usual Care
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2020-06-12): https://cdn.clinicaltrials.gov/large-docs/59/NCT03818659/Prot_SAP_ICF_000.pdf